CLINICAL TRIAL: NCT00897403
Title: Discovery of Candidate Biomarkers in Colon Cancer and Precancers Repository
Brief Title: Blood and Tissue Sample Collection for Future Colon Cancer Biomarker Studies in Patients Undergoing Colonoscopy
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Liebler, Adjunct Professor, Vanderbilt University Medical Center
Other Study IDs: CDR0000546530; P30CA068485 (NIH); VU-VICC-GI-0661; VU-VICC-IRB-061096
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer; Health Status Unknown
Keywords: colon cancer; health status unknown
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: biologic sample preservation procedure
Procedure: diagnostic colonoscopy

SUMMARY:
RATIONALE: Collecting and storing samples of blood and tissue from patients undergoing colonoscopy to study in the laboratory may help doctors learn more about colon cancer and identify biomarkers related to colon cancer in the future.

PURPOSE: This laboratory study is collecting blood and tissue samples for future colon cancer biomarker studies in patients undergoing colonoscopy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Collect blood and tissue samples (including polyps, abnormal growths, cancer, and normal tissue) from patients undergoing colonoscopy.

OUTLINE: Patients undergo blood and tissue sample collection during colonoscopy. Samples are stored for future biomarker proteomic profiling.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Scheduled for colonoscopy as routine screening or for a specific problem

PATIENT CHARACTERISTICS:

* Not pregnant

PRIOR CONCURRENT THERAPY:

* No concurrent participation in a clinical trial to treat cancer or prevent cancer recurrence

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for colonoscopy either as routine screening or for a specific problem.
Sampling Method: Non-Probability Sample
Enrollment: 6446 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Collection of blood and tissue | Pre-op & during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Liebler, PhD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Dan Rudy Cancer Center at Saint Thomas Hospital, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee